CLINICAL TRIAL: NCT00753727
Title: A Phase IB/II Study of Sunitinib in Combination With Neoadjuvant Radiation in Patients With Resectable Soft-tissue Sarcoma
Brief Title: Sunitinib and Radiation in Patients With Resectable Soft-tissue Sarcoma
Acronym: SUNXRT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Australasian Sarcoma Study Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Pfizer (Industry)
Responsible Party: Associate Professor David Thomas, Peter MacCallum Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSG01
Record Dates: First submitted 2008-09-14; First posted 2008-09-16 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-12

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue; Sarcoma; Sunitinib; neoadjuvant; radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Sunitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib dose 50 mg/day orally for 2 weeks prior to radiotherapy. Treatment Dose Levels during radiotherapy: Dose level 0: Sunitinib 50mg/day for 2 weeks prior to radiotherapy, followed by 25mg/day given concurrently with radiotherapy; Dose level 1: Sunitinib 50mg/day for 2 weeks prior to radiotherapy, followed by 37.5mg/day given concurrently with radiotherapy; Dose level -1: Sunitinib 37.5mg/day for 2 weeks prior to radiotherapy, followed by 37.5mg/day given concurrently with radiotherapy. Dose escalation/de-escalation: first 6 patients will be accrued at dose level 0. The dose levels at which subsequent patients will be accrued will be determined using a dose modification schedule.
  Other Names: Sutent
Radiation: Radiotherapy — Preoperative radiotherapy consisting of external beam radiotherapy at a dose of 50.4 Gy given in 28 fractions, five days a week, over five weeks and 3 days to the planning target volume.

SUMMARY:
This research is being done with the aim of developing a more effective treatment than standard radiotherapy and surgery alone. Although standard treatment is frequently successful, some patients do not respond well to this treatment. Low oxygen levels in tumours, which may be a particular problem with sarcomas, are thought to be one factor that contributes to failure of radiotherapy. Sunitinib is a new drug that is active against cells with low oxygen levels. The combination of sunitinib and radiotherapy has shown promising results in other cancers. The purpose of this study is to find out whether treatment with a new drug, sunitinib, can increase the effectiveness of radiotherapy at killing cancer cells; to test the safety of the combination of sunitinib and radiotherapy.

DETAILED DESCRIPTION:
The presence of hypoxia has been documented in soft-tissue sarcomas, where it may contribute to radioresistance. Combinations of radiosensitisers such as ifosfamide and doxorubicin with radiotherapy have demonstrated promise in sarcomas, but with significant toxicity.

The rationale for this study is based on:

* the frequency of hypoxia in soft-tissue sarcomas
* the importance of radiotherapy in neoadjuvant treatment of soft-tissue sarcomas
* targeting hypoxic vasculature with sunitinib
* the single agent activity of sunitinib in soft-tissue sarcomas. This study will assess the feasibility and tolerability of the combination of sunitinib with standard preoperative radiotherapy. The surrogate endpoints of tumor necrosis and functional and RECIST imaging response will provide early evidence of response rate. Toxicities will be assessed both during chemoradiation and following surgery. The impact of treatment on the hypoxic component of the tumor will be investigated with F18 azamycin arabinoside PET scans.

Because the combination of sunitinib and radiotherapy has not been studied before, we propose a phase Ib design with dose reductions in the event of excessive toxicity. Sunitinib treatment will precede the commencement of radiotherapy by 2 weeks because there is preclinical evidence that priming the tumor vasculature may increase synergy with radiotherapy, and because sunitinib may have single agent activity in sarcomas, including measurable effects on tumor vasculature. Because it is anticipated that the likelihood of complications attributable to the combination of sunitinib and radiotherapy will be small, the starting dose of sunitinib will be 50mg/day for the two week lead-in period and then 25mg for 5 weeks with concurrent radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed soft-tissue sarcoma suitable for neoadjuvant radiotherapy and surgery
* minimum age 16 years
* ECOG performance status =1
* life expectancy of greater than 6 months
* patients must have normal organ and marrow function
* no evidence of a bleeding or thrombotic tendency, and no evidence of arterial or venous thrombosis
* not pregnant or breastfeeding
* the ability to give written informed consent.

Exclusion Criteria:

* Soft-tissue sarcoma located in sites where radiotherapy is associated with significant exposure of abdominal viscera
* patients with other invasive malignancies, with the exception of non-melanoma skin cancer, in the last 5 years
* patients receiving any other therapeutic investigational agents
* patients who are receiving concurrent treatment with any other anti-cancer therapy
* evidence of distant metastases
* uncontrolled intercurrent illness
* patients who are pregnant or breast feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum dose of sunitinib at which the combination of sunitinib and radiotherapy pre-operatively is safe and tolerable. | Baseline; post-2 weeks sunitinib only administration; post-sunitinib and radiotherapy combination treatment; 12 weeks post-surgery

SECONDARY OUTCOMES:
To estimate response rates for the combination of sunitinib and radiotherapy. | Baseline; post-2 weeks sunitinib only administration; post-sunitinib and radiotherapy combination treatment; and at surgery

CONTACTS AND LOCATIONS:
Overall Officials: David Thomas, MB BS PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia